CLINICAL TRIAL: NCT01486342
Title: Positron Emission Tomography With [18F]Fluorodeoxyglucose in Patients at Risk for Acute Lung Injury
Brief Title: PET Imaging in Patients at Risk for Acute Lung Injury
Acronym: PET-ALI
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Brian Fuller, Assistant Professor of Anesthesiology and Emergency Medicine, Washington University School of Medicine
Other Study IDs: 201105122
Record Dates: First submitted 2011-11-21; First posted 2011-12-06 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Acute Lung Injury; Early Pulmonary Neutrophilic Inflammation
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Mechanically ventilated patients without acute lung injury and lung injury prediction score < 4
  Interventions: Radiation: PET-CT scan

INTERVENTIONS:
Radiation: PET-CT scan — PET-CT imaging with [18F]FDG will be performed within 24 hours of admission to the ICU. All patients imaged will be those remaining on mechanical ventilation at the time of PET imaging.
  A low-dose CT scan (50 effective mAs) will be obtained with placement of the participant such that the lungs are centered within the field of view. After completing the transmission scan, 10 mCi of [18F]FDG will be injected intravenously at the start of a 60-minute dynamic scan acquisition and the intravenous (IV) catheter flushed with 10 ml saline. Imaging will be obtained with the following framing schedule: 24 5-sec, 6 3-minute and 8 5-minute frames.

SUMMARY:
Despite decades of research, the mortality in acute lung injury remains very high and treatment options are very limited. Given these facts, the best treatment modality may be in prevention of this lethal syndrome.

Historically, imaging has played a crucial role in understanding ALI. The appearance of chest radiography is one of the consensus criteria in defining ALI, and commuted tomography (CT) scans further advanced the understanding of the pathoanatomy of ALI. While valuable, these imaging modalities are nonspecific and do not incorporate functional cellular physiology.

PET imaging measures concentrations of radioisotopes in the body. By embedding in, but not altering molecules, the natural fate of these tracers can be studied with PET imaging. Advances in the understanding of ALI include blood flow distribution, as well as the response to alveolar recruitment maneuvers and prone positioning. Not all patients who are receiving mechanical ventilation develop ALI. Inflammation in the lungs is known to play a key early role in the development and progression of ALI. Secondary to inflammation, the lungs develop edema and do not exchange oxygen as well. This early inflammation is in part driven by a specific type of immune cell called the neutrophil. These cells seem to travel and become sequestered in the lung- they are "recruited" to the lung during this inflammatory stage. When there, these neutrophils release inflammatory substances which are integral in the development of ALI. Neutrophils use primarily glucose as a fuel source. The radio isotope [18F]Fluorodeoxyglucose (FDG)is a glucose analog and therefore taken up/ingested by the neutrophils as a part of their normal metabolism. Because of this fact, positron emission tomography (PET) using the radio isotope [18F]FDG is a highly sensitive marker to look at the recruitment of neutrophils to the lung, therefore quantifying the degree of pulmonary inflammation prior to the development of ALI.

The investigators seek to examine the relationship of pulmonary inflammation in patients at risk for ALI, but without clinical evidence of the syndrome. The investigators seek to enroll ten patients in a pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (age ≥ 18) presenting to the SICU after ≥ 5 hours of mechanical ventilation in the OR or ED, without clinical evidence of ALI, and LIPS > 4 or < 4.
* Able to be positioned supine within the PET/CT scanner for ~1.25 hours
* Has legally authorized representative (LAR) available and willing to give informed consent, or is able to give informed consent prior to initiation of mechanical ventilation
* BMI < 35

Exclusion Criteria:

* Established ALI by accepted clinical criteria.
* Organ transplant recipient
* Treatment with immunosuppressive/immune-modulating medications
* Current corticosteroid treatment
* Chronic pulmonary or nonpulmonary inflammatory diseases
* Inability to safely travel out of the SICU (as established by regular safety screening criteria). Patient is placed in the supine position for a minimum of 30 minutes, and on mechanical ventilator settings that will be in place for the duration of the FDG-PET study. The patient is deemed unsafe for travel if oxygen requirement increases or any hemodynamic instability ensues (such as increasing vasopressor requirements).
* Glucose level > 150 mg/dl at time of PET scan
* Pregnancy (confirmed by qualitative urine hCG pregnancy test)
* Lactation
* Presence of implanted electronic medical device
* Enrollment in another research study of an investigational drug
* Prior research-related radiation exposure within the past year such that participation in this study would result in exposures that exceed the limits as defined by the FDA RDRC regulations (21 CFR 361.1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients without acute lung injury
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The influx constant (Ki) of FDG uptake | 3 days
  The influx constant describes the rate of FDG uptake and represents pulmonary inflammation

SECONDARY OUTCOMES:
Correlation of the influx constant (Ki) with lung injury prediction score | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Brian Fuller, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States